CLINICAL TRIAL: NCT04851483
Title: Characterization of Single Dose Bioavailability of Two Novel Formulations of BAY 2328065 in Healthy Male Participants Including Dose Proportionality of One Formulation and Investigation of Safety, Tolerability and Pharmacokinetics of Multiple Dose Administration in Healthy Female Participants
Brief Title: A Trial to Learn What Happens to Different Medicinal Forms of BAY2328065 When They Enter the Body and How Safe They Are in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20568; 2020-005497-96 (EudraCT Number)
Record Dates: First submitted 2021-04-16; First posted 2021-04-20 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: * Study Groups 1 and 2 using a fixed sequence parallel group design
  * Study Group 3 using a fixed sequence design
  * Study Group 4 using a placebo-controlled parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Study Groups 1 and 2: open-label
  * Study Group 3: open-label
  * Study Group 4: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1_BAY2328065 _male participants (Experimental): Approximately 6 participants will be randomly assigned to one of the 2 study intervention sequences (Group 1 or Group 2).
  Interventions: Drug: BAY2328065
- Group 2_BAY2328065 _male participants (Experimental): Approximately 6 participants will be randomly assigned to one of the 2 study intervention sequences (Group 1 or Group 2).
  Interventions: Drug: BAY2328065
- Group 3_BAY2328065 _male participants (Experimental): Approximately 8 participants will be assigned to the study intervention with one fixed sequence.
  Interventions: Drug: BAY2328065
- Group 4_BAY2328065 _female participants (Experimental): Approximately 9 participants will be randomly assigned to receive BAY2328065.
  Interventions: Drug: BAY2328065
- Group 4_Placebo _female participants (Placebo Comparator): Approximately 3 participants will be randomly assigned to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY2328065 — Solid Form, Oral administration.
  Arms: Group 1_BAY2328065 _male participants; Group 2_BAY2328065 _male participants; Group 3_BAY2328065 _male participants; Group 4_BAY2328065 _female participants
Drug: Placebo — Matching placebo of BAY2328065.
  Arms: Group 4_Placebo _female participants

SUMMARY:
Researchers are looking for a different way to treat women with a condition in which tissue that normally lines the uterus grows outside the uterus. This condition is called endometriosis. Before a treatment is available to all patients, researchers study it in clinical trials to better understand its safety and what happens to it in the body.

BAY2328065 is being developed to help treat women who have endometriosis. Women with endometriosis often have very painful menstrual periods, as well as pain in the pelvic area which is not related to menstrual periods and pain during intercourse. Many women with endometriosis may also have problems becoming pregnant. The trial treatment, BAY2328065, works by blocking a certain protein that causes pain and swelling of the tissue and is thought to play a role in endometriosis.

In this trial, the researchers want to compare what happens to different medicinal forms of BAY2328065 in the body. They also want to learn if eating a meal affects what happens to BAY2328065 in the body.

This trial will include about 32 men and women who are aged 18 to 55. There will be 4 groups of participants in this trial. The participants in Groups 1, 2, and 3 will be men. The participants in Group 4 will be women. There will be 3 treatment courses to the trial for Groups 1, 2 and 3 and 1 treatment course for Group 4.

During the trial, the participants in Groups 1, 2, and 3 will stay at the trial site for 15 days (3 times 5 days with times in between during which they stay at home). The participants in Group 4 will stay at the trial site for 16 days continuously. But, the trial will last about 6 weeks for the participants in Groups 1, 2, and 3. The trial will last about 9 weeks for the participants in Group 4.

All of the participants in Groups 1 and 2 will take the different medicinal forms of BAY2328065, with and without food. All of the participants in Groups 1 and 2 will take dose "2" of BAY2328065 in all 3 treatment courses. In Group 1, they will take BAY2328065 one time each during the following treatment courses:

* A medicinal form of BAY2328065 without food in treatment course 1, then
* A medicinal form of BAY2328065 differing from the one used in treatment course 1 without food in treatment course 2, then
* The medicinal form of BAY2328065 used in treatment course 1 with food in treatment course 3 The participants in Group 2 will do the same, but they will take each form of BAY2328065 in a different order. Information gathered from Group 1 and 2 will help the researchers learn which form of BAY2328065 will be most suited to give to the participants in Groups 3 and 4.

The participants in Group 3 will take 3 different doses of BAY2328065 with food in each treatment course. They will take one time each during the following treatment courses:

* Single administration of dose "1" in treatment course 1, then
* Single administration of dose "2" in treatment course 2, then
* Single administration of dose "3" in treatment course 3 This will help the researchers learn the safest dose to give to the participants in treatment course 4.

The participants in Group 4 will either take dose "3" or "2" of BAY2328065 based on the results of treatment course 3, or a placebo. A placebo looks like a treatment but does not have any medicine in it. All of the participants will take either:

* Multiple administrations of dose "3" of BAY2328065 or dose "2" of BAY2328065, OR
* the placebo The participants will take BAY2328065 or placebo over 12 days without food.

The doctors/ healthcare staff will:

* take blood and collect urine samples
* check the participants' heart health

The participants will:

* answer questions about how they are feeling
* say if they have any medical problems
* say if they have taken any medications

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent
* Participants must be overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, ECG, blood pressure and heart rate
* Confirmation of the subject's health insurance coverage prior to the first screening examination/visit
* Body mass index (BMI) within the range 18 and 30 kg/m^2 (inclusive)
* Male participants who are sexually active and female participants of childbearing potential must use one of the methods of contraception described in this protocol

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal
* Relevant diseases within the last 4 weeks prior to start of the first study intervention
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Existing chronic diseases as specified in protocol
* Regular use of therapeutic or recreational drugs
* Suspicion of drug or alcohol abuse
* Smoking equal or more than 10 cigarettes/day
* History of COVID-19; contact with SARS-CoV-2 positive persons or COVID-19 patients within the last 4 weeks prior admission to the ward or positive SARS-CoV-2 viral RNA test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAE) | From first administration of study intervention up to 30 days after end of treatment with study intervention
Severity of treatment-emergent adverse events (TEAEs) | From first administration of study intervention up to 30 days after end of treatment with study intervention
AUC of BAY2328065 | From dosing up to 72 hours
  AUC: area under the concentration vs. time curve from zero to infinity after single (first) dose
Cmax of BAY2328065 | From dosing up to 72 hours
  Cmax: maximum observed drug concentration in measured matrix after single dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.